CLINICAL TRIAL: NCT01059422
Title: Efficacy and Safety of an Initial Regimen Raltegravir (RAL) + Lamivudine/Abacavir Fixed-Dose Combination (3TC/ABC FDC) for 48 Weeks in ART- naïve, HIV/TB Co-Infected Adult Subjects Receiving Rifabutin-containing, 1-line Anti-TB Therapy
Brief Title: Raltegravir + Lamivudine/Abacavir in HIV/Tuberculosis Co-Infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central Institute of Epidemiology, Moscow, Russia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Vadim Pokrovsky, Professor, Central Institute of Epidemiology, Moscow, Russia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAL/ABC/3TC - HIV/TB
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: HIV Infections; Tuberculosis
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — Raltegravir Potassium; abacavir; Lamivudine; abacavir, lamivudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Raltegravir; Abacavir/Lamivudine (Experimental): Raltegravir: 400 mg twice daily Abacavir/Lamivudine fixed-dose combination: 600mg/300mg once daily
  Interventions: Drug: Raltegravir; Abacavir/Lamivudine

INTERVENTIONS:
Drug: Raltegravir; Abacavir/Lamivudine — Raltegravir: 400 mg twice daily Abacavir/Lamivudine fixed-dose combination: 600mg/300mg once daily
  Other Names: Isentress®; Epzicom®

SUMMARY:
The study will investigate whether combination antiretroviral therapy of raltegravir and 3TC/ABC is effective and safe to use in tuberculosis (TB)/HIV co-infected adults receiving rifabutin-containing, first-line antituberculous treatment.

Hypothesis:Combination antiretroviral therapy of raltegravir and 3TC/ABC and is effective and safe to use in tuberculosis (TB)/HIV co-infected adults receiving rifabutin-based first-line antituberculous treatment.

DETAILED DESCRIPTION:
This is a phase IIIB/IV, open-label, multi-center, single-arm descriptive pilot study of the efficacy and safety of RAL BID in combination with ABC/3TC QD in antiretroviral-naïve HIV-1 infected individuals with a presumptive or confirmed diagnosis of tuberculosis, without planned comparative analyses.

A goal of 40 subjects will be enrolled from 3 sites in the Russian Federation, including in our site, and receive RAL BID + 3TC/ABC QD for 48 weeks.

This study will include screening, treatment and follow-up periods. Screening period up to 28 days includes initial visits at Day -28 (screening) and Day -14 (switch to rifabutin). The second visit will be required if patient is initially on rifampin-based TB regimen that will need to be switched to rifabutin-based regimen.

Patients receiving rifampin-containing TB therapy will be switched to rifabutin (300 mg daily) a minimum of 14 days prior to initiation of antiretroviral therapy. Patients must not have received more than 45 days of tuberculosis therapy.

Treatment period from Day 1 to Week 48 includes 7 visits and a follow-up period (2-4 weeks after the Week 48 visit or Withdrawal visit) includes one visit for resolution of ongoing AEs (adverse events) and new SAEs (serious adverse events). Patients will therefore have 10 scheduled assessments: screening (Day -28; Day -14), baseline (Day 1), Weeks 4, 8, 12, 24, 36, and 48, and follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* ART-naïve HIV infected patients
* Plasma HIV-1 RNA >1,000 copies/mL at screening
* CD4 cells 100-350 cells/mm3
* Have presumptive or confirmed diagnosis of Mycobacterium tuberculosis infection
* Receiving first-line antituberculosis treatment
* Documented negative results for the presence of HLA-B*5701 allele

Exclusion Criteria:

* Pregnancy and Breastfeeding
* Known allergy/sensitivity to study drugs or their formulations
* A condition (including but not limited to active alcohol or drug use) that, in the opinion of the investigator, may interfere with patient adherence or safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-10; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with plasma HIV-1 RNA <50 copies/ml by the Time to Loss of Virologic Response (TLOVR) algorithm | 48 week
  It's included in the primary outcome measure title.

CONTACTS AND LOCATIONS:
Overall Officials: Vadim V. Pokrovsky, PhD, Principal Investigator — Central Research Institute of Epidemiology
Locations (1):
- Central Research Institute of Epidemiology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No